CLINICAL TRIAL: NCT03012789
Title: Diagnosis of Neuroendocrine Neoplasms and Assessment of Response to Surgery by Means of Measurement of Gene Transcripts in Blood
Brief Title: Surgical Intervention and the NETest
Acronym: NETest_Sx
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wren Laboratories LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Surgery_NETest
Record Dates: First submitted 2016-12-06; First posted 2017-01-06 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Neuroendocrine Tumor; Gastroenteropancreatic
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post Surgery (Other)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgical excision

SUMMARY:
The purpose of this study is to evaluate the effect of different surgical resections (R0, R1, R2) on circulating NET transcripts (PCR score or NETest). A drop in circulating NET levels will be correlated with surgical excision. Secondly, variation of circulating NET transcripts will be correlated to NET recurrence to test whether this analysis may constitute an early predictive marker of disease relapse.

DETAILED DESCRIPTION:
Biomarker-based tools that can accurately predict gastroenteropancreatic neuroendocrine tumor (GEP-NET) treatment response and tumor recurrence are currently not available. Circulating biomarkers that are associated with GEP-NETs are limited to measurements of plasma chromogranin A (CgA). The investigators have developed a PCR-based tool to quantitate (score) the circulating GEP-NET molecular signature ("liquid" biopsy) with high sensitivity and specificity. This signature can identify all types of GEP-NETs including small (1cm) non-metastatic tumors, is significantly reduced after tumor debulking and is decreased following surgical "cure". Elevated post-surgical scores are associated with tumor recurrence within 6 months in ~40% of cases. Current NET treatment protocols are associated with tumor recurrence (progression free survival) ranging from 5-18 months. The majority of patients will experience a relapse within 18 months irrespective of the treatment approach. The investigators hypothesize that a PCR measurement of circulating NET mRNA can accurately predict the extent of surgical resection (tumor removal) and elevated scores can predict tumor relapse before this occurs. This biomarker protocol seeks to test this hypothesis and evaluate whether changes in plasma CgA are as effective in predicting resection and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, well differentiated (G1, G2 or G3), local and advanced (metastatic), neuroendocrine tumor of gastro-enteropancreatic origin.
* Treatment-naïve as well as patients who have received previous therapies.
* Patients currently on LAR with clinically stable disease.
* CT or MRI documentation of disease.
* WHO performance status ≤2.

Exclusion Criteria:

* Known history of HIV seropositivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Biomarker prediction of tumor recurrence | 24 months
  Analysis of the alterations in the biomarker levels (from post-surgical levels, i.e., month 1) will be utilized to establish when the disease status has altered; a sustained increase in score will be recorded and compared with imaging to assess whether this is associated with disease progression/recurrence.

SECONDARY OUTCOMES:
Biomarkers and clinical symptomatology | 24 months
  Biomarker scores will be compared to the frequency of clinical symptoms, specifically flushing, to assess whether there is a relationship.
Biomarkers and clinical symptomatology | 24 months
  Biomarker scores will be compared to the frequency of clinical symptoms, specifically diarrhea, to assess whether there is a relationship.

OTHER OUTCOMES:
Alteration in biomarkers and tumor removal | 24 months
  Analysis of the change in biomarker scores (from baseline to post-surgical levels at 1 month) will be utilized to establish the strength of the relationship between the biomarker and volume of tumor removed (cm3).

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital IRCCS, Milan, Italy

REFERENCES:
- [Result] Modlin IM, Frilling A, Salem RR, Alaimo D, Drymousis P, Wasan HS, Callahan S, Faiz O, Weng L, Teixeira N, Bodei L, Drozdov I, Kidd M. Blood measurement of neuroendocrine gene transcripts defines the effectiveness of operative resection and ablation strategies. Surgery. 2016 Jan;159(1):336-47. doi: 10.1016/j.surg.2015.06.056. Epub 2015 Oct 9. PMID 26456125
- [Result] Modlin IM, Kidd M, Bodei L, Drozdov I, Aslanian H. The clinical utility of a novel blood-based multi-transcriptome assay for the diagnosis of neuroendocrine tumors of the gastrointestinal tract. Am J Gastroenterol. 2015 Aug;110(8):1223-32. doi: 10.1038/ajg.2015.160. Epub 2015 Jun 2. PMID 26032155
- [Result] Oberg K, Modlin IM, De Herder W, Pavel M, Klimstra D, Frilling A, Metz DC, Heaney A, Kwekkeboom D, Strosberg J, Meyer T, Moss SF, Washington K, Wolin E, Liu E, Goldenring J. Consensus on biomarkers for neuroendocrine tumour disease. Lancet Oncol. 2015 Sep;16(9):e435-e446. doi: 10.1016/S1470-2045(15)00186-2. PMID 26370353